CLINICAL TRIAL: NCT01565707
Title: A Phase 3, Double-Blind, Randomized, Multi-center, Placebo-Controlled Sequential Dose Titration Study to Assess Efficacy, Safety and Population Pharmacokinetics of Solifenacin Succinate Suspension in Pediatric Subjects From 5 to Less Than 18 Years of Age With Overactive Bladder (OAB)
Brief Title: A Study to Investigate How Effective and Safe Solifenacin Succinate Suspension is in Treating Children/Adolescents Aged 5 to Less Than 18 Years With Symptoms of Overactive Bladder (OAB) Compared to a Non-active Drug
Acronym: LION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-CL-076; 2011-002066-20 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Pediatric; Solifenacin succinate suspension; Phase 3; Pharmacokinetics; Overactive bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Children (Placebo Comparator): Children aged 5 to 11 years received matching placebo suspension once a day for 12 weeks.
  Interventions: Drug: Placebo; Behavioral: Urotherapy
- Solifenacin Succinate Suspension Children (Experimental): Children aged 5 to 11 years received solifenacin succinate suspension once a day for 12 weeks. The initial dose started with pediatric equivalent dose (PED) of 5 mg (PED5) based on weight and was titrated up or down to reach the optimal dose. The minimum dose was PED2.5, and the maximum dose was PED10.
  Interventions: Drug: Solifenacin Succinate Suspension; Behavioral: Urotherapy
- Placebo Adolescents (Placebo Comparator): Adolescents aged 12 to 17 years received matching placebo suspension once a day for 12 weeks.
  Interventions: Drug: Placebo; Behavioral: Urotherapy
- Solifenacin Succinate Suspension Adolescents (Placebo Comparator): Adolescents aged 12 to 17 years received solifenacin succinate suspension once a day for 12 weeks. The initial dose started with pediatric equivalent dose (PED) of 5 mg (PED5) based on weight and was titrated up or down to reach the optimal dose. The minimum dose was PED2.5, and the maximum dose was PED10.
  Interventions: Drug: Solifenacin Succinate Suspension; Behavioral: Urotherapy

INTERVENTIONS:
Drug: Solifenacin Succinate Suspension — Children aged 5 to 11 years and adolescents aged 12 to 17 years received solifenacin succinate liquid suspension once a day orally via syringe for 12 weeks along with non interventional diary assisted urotherapy consisting of overactive bladder (OAB) information, awareness, instruction, life-style advice and documentation of voiding habits and symptoms for OAB. The initial dose started with the equivalent of 5 mg in adults, referred to as pediatric equivalent dose (PED) of 5 mg (PED5), based on body weight for three weeks and was titrated up or down in up to three titration steps of three weeks each to reach the optimal dose. Titration up or down could lead to weight-based doses equivalent to doses in adults of 2.5 mg, 5 mg, 7.5 mg or 10 mg once daily and were referred to as PED2.5, PED5, PED7.5 and PED10. The minimum dose was PED2.5, and the maximum dose was PED10. The decision to titrate up or down was made by the investigator using information from the 7 day patient diary.
  Other Names: YM905
  Arms: Solifenacin Succinate Suspension Adolescents; Solifenacin Succinate Suspension Children
Drug: Placebo — Children aged 5 to 11 years and adolescents aged 12 to 17 years received matching placebo liquid suspension once a day orally via syringe for 12 weeks along with non interventional diary assisted urotherapy consisting of overactive bladder (OAB) information, awareness, instruction, life-style advice and documentation of voiding habits and symptoms for OAB. The initial dose started with the equivalent of 5 mg in adults, referred to as pediatric equivalent dose (PED) of 5 mg (PED5), based on body weight for three weeks and was titrated up or down in up to three titration steps of three weeks each to reach the optimal dose. Titration up or down could lead to weight-based doses equivalent to doses in adults of 2.5 mg, 5 mg, 7.5 mg or 10 mg once daily and were referred to as PED2.5, PED5, PED7.5 and PED10. The minimum dose was PED2.5, and the maximum dose was PED10. The decision to titrate up or down was made by the investigator using information from the 7 day patient diary.
  Arms: Placebo Adolescents; Placebo Children
Behavioral: Urotherapy — Non interventional diary assisted urotherapy consisting of overactive bladder (OAB) information, awareness, instruction, life-style advice and documentation of voiding habits and symptoms for OAB.
  Other Names: Bladder training

SUMMARY:
Solifenacin succinate as a tablet formulation is already on the market for the treatment of symptoms of overactive bladder in adults. For the use in children and adolescent patients a new formulation of solifenacin has been developed.

This study investigated the effect and safety of solifenacin succinate liquid suspension compared to a non-active drug (placebo) over a 12-week period. The 2 weeks prior to the double blind period was a single-blind placebo run-in period in combination with behavioral urotherapy (Non-interventional diary assisted urotherapy consisting of overactive bladder (OAB) information, awareness, instruction, life-style advice and documentation of voiding habits and symptoms for OAB), followed by a 12 week daily treatment period. The study also investigated how well solifenacin succinate suspension is taken-up by the body and how long it stays in the body during this time.

ELIGIBILITY:
Main Inclusion Criteria:

* Written Informed Consent has been obtained
* OAB (symptoms of urgency) according to International Children's Continence Society (ICCS) criteria
* Daytime incontinence with at least 4 or more episodes of incontinence confirmed by 7 day participant diary

Main Exclusion Criteria:

* Daily voiding frequency less than 5
* Extraordinary daytime urinary frequency according to the International Children's Continence Society (ICCS) definition
* Uroflow indicative of pathology other than OAB
* Maximum voided volume (morning volume excluded) > expected bladder capacity for age [(age +1) x 30] in ml or a maximum voided volume (morning volume excluded) above 390 ml
* Post Void Residual (PVR) > 20 ml
* Monosymptomatic enuresis
* Polyuria defined as > 75 ml/kg/b.w./24 hours
* Dysfunctional voiding
* Congenital anomalies affecting lower urinary tract function
* Current constipation
* Current Urinary Tract Infection (UTI)
* Catheterization within 2 weeks prior to screening

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2014-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (46):
- United States (2):
  - Site: 1006, Shreveport, Louisiana
  - Site: 1015, Albany, New York
- Belgium (7):
  - Site: 3202, Antwerp
  - Site: 3209, Antwerp
  - Site: 3208, Charleroi
  - Site: 3201, Ghent
  - Site: 3203, Ghent
  - Site: 3204, Kortrijk
  - Site: 3205, Leuven
- Brazil (2):
  - Site: 5507, Campinas
  - Site: 5506, Curitiba
- Canada (2):
  - Site: 1005, Hamilton
  - Site: 1001, Québec
- Denmark (4):
  - Site: 4503, Aalborg
  - Site: 4501, Aarhus N
  - Site: 4502, Kolding
  - Site: 4504, Køge
- Mexico (2):
  - Site: 5202, Mexico City
  - Site: 5205, Mexico City
- Norway (2):
  - Site: 4701, Bergen
  - Site: 4702, Trondheim
- Site: 6301, Quezon City, Philippines
- Poland (4):
  - Site: 4805, Gdansk
  - Site: 4803, Gdansk
  - Site: 4804, Lubin
  - Site: 4801, Warsaw
- Serbia and Montenegro (2):
  - Site: 3810, Belgrade
  - Site: 3812, Novi Sad
- Site: 2703, Cape Town, South Africa
- South Korea (5):
  - Site:8203, Daegu
  - Site: 8206, Incheon
  - Site: 8207, Seoul
  - Site: 8201, Seoul
  - Site:8202, Seoul
- Sweden (5):
  - Site: 4606, Gothenburg
  - Site: 4601, Jönköping
  - Site: 4603, Skövde
  - Site: 4602, Stockholm
  - Site: 4605, Umeå
- Turkey (Türkiye) (2):
  - Site: 9001, Ankara
  - Site: 9002, Izmir
- Ukraine (3):
  - Site: 3853, Dnipropetrovsk
  - Site: 3854, Kharkiv
  - Site: 3850, Kiev
- United Kingdom (2):
  - Site: 4403, Leeds
  - Site: 4401, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Tannenbaum S, den Adel M, Krauwinkel W, Meijer J, Hollestein-Havelaar A, Verheggen F, Newgreen D. Pharmacokinetics of solifenacin in pediatric populations with overactive bladder or neurogenic detrusor overactivity. Pharmacol Res Perspect. 2020 Dec;8(6):e00684. doi: 10.1002/prp2.684. PMID 33231929
- [Derived] Snijder R, Bosman B, Stroosma O, Agema M. Relationship between mean volume voided and incontinence in children with overactive bladder treated with solifenacin: post hoc analysis of a phase 3 randomised clinical trial. Eur J Pediatr. 2020 Oct;179(10):1523-1528. doi: 10.1007/s00431-020-03635-2. Epub 2020 Apr 1. PMID 32239291
- [Derived] Newgreen D, Bosman B, Hollestein-Havelaar A, Dahler E, Besuyen R, Sawyer W, Bolduc S, Rittig S. Solifenacin in Children and Adolescents with Overactive Bladder: Results of a Phase 3 Randomised Clinical Trial. Eur Urol. 2017 Mar;71(3):483-490. doi: 10.1016/j.eururo.2016.08.061. Epub 2016 Sep 28. PMID 27687820
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=239

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of male and female children (5 to 11 years old) and adolescents (12 to 17 years old) with overactive bladder (OAB).
Pre-assignment Details: Subjects received 4 weeks of urotherapy (standard first line therapy for pediatric OAB patients). Two weeks after start of urotherapy a single-blind 2-week placebo run-in period began. After run-in period eligible subjects were randomized to 12 weeks of double-blind treatment (solifenacin succinate suspension or placebo) and continued urotherapy.
Period: Overall Study
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Started | 75 | 73 | 19 | 22
Treated | 73 | 73 | 19 | 22
Completed | 66 | 65 | 16 | 17
Not Completed | 9 | 8 | 3 | 5
Not completed — Adverse Event | 1 | 6 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1
Not completed — Randomized but not evaluable | 2 | 0 | 0 | 0
Not completed — Miscellaneous | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline values provided are based on the Safety Analysis Set (SAF) population and the Full Analysis Set (FAS). Population analysis is defined within each baseline measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents | Total
Number analyzed (Participants) | 73 | 73 | 19 | 22 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] — Age values provided are for the Safety Analysis Set (SAF) population. The SAF consisted of all participants who received at least 1 dose of double-blind study medication and for whom any safety data were reported after first dose of study drug. The number of participants was 73; 73; 19; 22 per treatment arm.
  years
    Children | 7.4 (1.6) | 7.6 (1.6) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 7.5 (1.6)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 14.4 (1.9) | 14.2 (1.8) | 14.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — SAF population. The number of participants was 73; 73: 19; 22 per treatment arm.
  Participants
    Female | 35 | 44 | 16 | 17 | 112
    Male | 38 | 29 | 3 | 5 | 75
Race [Number; unit: Participants] — SAF population. The number of participants was 73; 73; 19; 22 per treatment arm.
  Participants
    White | 57 | 62 | 13 | 16 | 148
    Black/African American | 3 | 2 | 1 | 2 | 8
    Asian | 6 | 5 | 3 | 4 | 18
    American Indian/Alaskan Native | 3 | 4 | 2 | 0 | 9
    Other | 4 | 0 | 0 | 0 | 4
Ethnicity [Number; unit: Participants] — SAF population. The number of participants was 73; 73; 19; 22 per treatment arm.
  Participants
    Hispanic or Latino | 8 | 9 | 3 | 2 | 22
    Not Hispanic or Latino | 65 | 64 | 16 | 20 | 165
Mean Volume Voided (MVV) per Micturition [Mean (Standard Deviation); unit: mL] — Values for this baseline characteristic are based on the Full Analysis Set (FAS). The FAS consisted of all randomized patients that took at least 1 dose of double-blind study medication after randomization and provided a valid baseline and post baseline value for the primary efficacy endpoint. A micturition is any voluntary urination, excluding episodes of incontinence only. Micturitions voided volumes were recorded in a patient diary for any 2 days in the 7 day period prior to the baseline visit (referred to as "measuring days"). The number of participants was 70; 73; 19; 21 per arm.
  mL
    Children | 94.06 (38.12) | 96.88 (40.98) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 95.50 (39.50)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 169.06 (63.65) | 159.55 (61.21) | 164.07 (61.76)
Daytime Maximum Volume Voided (DMaxVV) Per Micturition [Mean (Standard Deviation); unit: mL] — FAS population. The mean DMaxVV was determined using the patient diary data recorded during two measuring days (i.e., days when the patient recorded the volume of each micturition) in the 7 days prior to the baseline visit. The DMaxVV is the largest (non-zero) volume recorded over both of the 2 measuring days in the diary (first morning void excluded). Daytime defined as time between waking up in the morning and going to bed later the same day. A micturition is any voluntary urination, excluding episodes of incontinence only. The number of participants was 70; 73; 19; 21 per treatment arm.
  mL
    Children | 141.43 (52.09) | 155.51 (70.66) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 148.62 (62.45)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 278.16 (119.21) | 252.38 (108.68) | 264.63 (113.08)
Mean Number of Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: incontinence episodes] — FAS population. The mean of the number of incontinence episodes was determined using diary data recorded by the participant in the 7 days prior to baseline visit. An incontinence episode is defined as an episode with any involuntary loss of urine. The number of participants was 70; 73; 19; 21 per treatment arm.
  incontinence episodes
    Children | 2.98 (2.63) | 2.46 (2.57) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 2.71 (2.60)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 2.81 (2.45) | 1.82 (1.66) | 2.29 (2.11)
Mean Number of Daytime Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: daytime incontinence episodes] — FAS population. The mean of the number of incontinence episodes was determined using diary data recorded by the participant in the 7 days prior to baseline visit. Daytime is defined as the time between waking up in the morning and going to bed later the same day. An incontinence episode is defined as an episode with any involuntary loss of urine. The number of participants was 70; 71; 19; 21 per treatment arm.
  daytime incontinence episodes
    Children | 2.54 (2.75) | 1.98 (3.24) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 2.26 (3.01)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 2.03 (2.18) | 1.50 (1.44) | 1.75 (1.83)
Mean Number of Nighttime Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: nighttime incontinence episodes] — FAS population. The mean of the number of incontinence episodes was determined using diary data recorded by the participant in the 7 days prior to baseline visit. An incontinence episode is defined as an episode with any involuntary loss of urine. Nighttime is defined as the time between going to bed and waking up the following morning. The number of participants was 70; 71; 19; 21 per treatment arm.
  nighttime incontinence episodes
    Children | 0.59 (0.47) | 0.70 (0.82) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 0.64 (0.67)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 0.39 (0.66) | 0.33 (0.40) | 0.36 (0.53)
Number of Dry (Incontinence-free) Days per 7 Days [Mean (Standard Deviation); unit: Dry Days] — FAS population. The mean of the number of dry days was determined using diary data recorded by the participant in the 7 days prior to baseline visit. The number of participants was 70; 73; 19; 21 per treatment arm.
  Dry Days
    Children | 0.5 (0.9) | 0.9 (1.6) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 0.7 (1.3)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 1.0 (1.0) | 1.5 (1.3) | 1.3 (1.2)
Number of Dry (Incontinence-free) Nights per 7 Days [Mean (Standard Deviation); unit: Dry Nights] — FAS population. The mean of the number of dry nights was determined using diary data recorded by the participant in the 7 days prior to baseline visit. The number of participants was 70; 73; 19; 21 per treatment arm.
  Dry Nights
    Children | 3.4 (3.0) | 3.1 (3.0) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 3.2 (3.0)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 5.6 (2.2) | 5.4 (2.2) | 5.5 (2.2)
Mean Number of Micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions] — FAS population. The mean of the number of micturitions was determined using diary data recorded by the participant in the 7 days prior to baseline visit. A micturition is any voluntary urination, excluding episodes of incontinence only. The number of participants was 70; 73; 19; 21 per treatment arm.
  micturitions
    Children | 8.26 (2.56) | 8.27 (3.01) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 8.27 (2.79)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 8.08 (3.82) | 7.52 (2.37) | 7.79 (3.11)
Mean Number of Daytime Micturitions per 24 Hours [Mean (Standard Deviation); unit: daytime micturitions] — FAS population. The mean of the number of micturitions was determined using diary data recorded by the participant in the 7 days prior to baseline visit. A micturition is any voluntary urination, excluding episodes of incontinence only. The number of participants was 70; 71; 19; 21 per treatment arm.
  daytime micturitions
    Children | 7.54 (3.14) | 8.00 (3.40) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 7.77 (3.27)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 6.79 (2.92) | 6.88 (2.14) | 6.84 (2.51)
Mean Number of Nighttime Micturitions per 24 Hours [Mean (Standard Deviation); unit: nighttime micturitions] — FAS population. The mean of the number of micturitions was determined using diary data recorded by the participant in the 7 days prior to baseline visit. A micturition is any voluntary urination, excluding episodes of incontinence only. The number of participants was 70; 71; 19; 21 per treatment arm.
  nighttime micturitions
    Children | 0.60 (0.78) | 0.56 (0.98) | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 0.58 (0.88)
    Adolescents | NA (NA) — Category not applicable to the arm. | NA (NA) — Category not applicable to the arm. | 0.61 (1.09) | 0.26 (0.41) | 0.43 (0.81)
Mean Number of Grade 3 or 4 Urgency Episodes per 24 Hours in Adolescents [Mean (Standard Deviation); unit: urgency episodes] — FAS population. Adolescent participants were asked to record the degree of urgency associated with each micturition and incontinence episode according to the Patient Perception of Intensity of Urgency Scale (PPIUS) scale (0 - no urgency, 1 - mild urgency, 2 - moderate urgency, 3 - severe urgency, 4 - urge incontinence). The mean number of grade 3 or 4 urgency episodes was determined using diary data recorded by the participant in the 7 days prior to baseline visit. The number of participants was N/A; N/A; 19; 20 per treatment arm.
  urgency episodes | NA (NA) — Baseline measure not applicable to the arm. | NA (NA) — Baseline measure not applicable to the arm. | 3.67 (4.15) | 2.42 (2.13) | 3.03 (3.29)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EoT) in Mean Volume Voided (MVV) Per Micturition
Description: The mean voided volume was calculated from the participant diary data recorded during two measuring days (i.e., those days when the participant recorded the volume of each micturition) in the 7 days prior to the baseline and end of treatment visits. The MVV is equal to the mean of the non-zero volumes recorded over the 2 measuring days. A micturition is any voluntary urination, excluding episodes of incontinence.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) consists of all randomized patients that took at least one dose of double-blind study medication after randomization and provided both valid baseline and post-baseline values for the primary efficacy endpoint. Missing values at EoT were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 73 | 19 | 21
mL | 13.4 (4.8) | 25.5 (4.8) | 6.9 (14.6) | 2.3 (14.0)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; The following hypotheses were tested at the 2-sided significance level 0.05: * H0: Change from baseline to EoT in mean MVV per micturition is the same for placebo and solifenacin succinate oral suspension * H1: Change from baseline to EoT in mean MVV per micturition is not the same for placebo and solifenacin succinate oral suspension; Test type: Superiority or Other; p = 0.046, ANCOVA; From an ANCOVA (analysis of covariance) model including treatment, geographic region & gender as fixed effects & the baseline value as a covariate; Adjusted Mean Difference = 12.1, 95% CI 2-sided [0.2 to 24.0], Standard Error of Mean 6.0
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = -4.7, 95% CI 2-sided [-36.7 to 27.4], Standard Error of Mean 15.7 — From an ANCOVA model including treatment, geographic region & gender as fixed effects & the baseline value as a covariate

2. Secondary Outcome: Change From Baseline to End of Treatment in Daytime Maximum Volume Voided (DMaxVV) Per Micturition
Description: The mean daytime maximum volume voided (DMaxVV) was determined using the participant diary data recorded during two measuring days (i.e., those days when the participant recorded the volume of each micturition) in the 7 days prior to the Baseline and end of treatment visits. The daytime maximum volume voided (DMaxVV) is the largest (non-zero) volume recorded over both of the 2 measuring days in the diary. The first morning void is excluded from the calculation. Daytime is defined as the time between waking up in the morning and going to bed later the same day. A micturition is any voluntary urination, excluding episodes of incontinence.
Time Frame: Baseline and Week 12
Population: The study analysis population for this endpoint consisted of the FAS population. Missing values at EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 73 | 19 | 21
mL | 11.3 (11.2) | 43.2 (11.1) | -8.4 (27.0) | -25.7 (26.3)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.024, ANCOVA; From an ANCOVA model including treatment, geographic region & gender as fixed effects & the baseline value as a covariate; Adjusted Mean Difference = 31.9, 95% CI 2-sided [4.3 to 59.5], Standard Error of Mean 13.9
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = -17.3, 95% CI 2-sided [-76.5 to 41.9], Standard Error of Mean 29.1 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode is defined as an episode with any involuntary loss of urine. The mean number of incontinence episodes was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 73 | 19 | 21
incontinence episodes | -1.2 (0.2) | -1.1 (0.2) | -0.7 (0.4) | -0.6 (0.4)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.763, ANCOVA — P-value is from a rank ANCOVA analysis stratified by geographic region; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-0.8 to 1.0], Standard Error of Mean 0.4 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Daytime Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. An incontinence episode is defined as an episode with any involuntary loss of urine. Daytime is defined as the time between waking up in the morning and going to bed later the same day.
Time Frame: Baseline and Week 12
Population: Full analysis set including patients for whom data were available. Missing values at EoT were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: daytime incontinence episodes
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 71 | 19 | 21
daytime incontinence episodes | -1.1 (0.2) | -1.2 (0.2) | -0.2 (0.4) | -0.8 (0.4)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.402, ANCOVA — P-value is from a rank ANCOVA analysis stratified by geographic region; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = -0.6, 95% CI 2-sided [-1.5 to 0.4], Standard Error of Mean 0.5 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Nighttime Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. An incontinence episode is defined as an episode with any involuntary loss of urine. Nighttime is defined as the time between going to bed and waking up the following morning.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nighttime incontinence episodes
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 71 | 19 | 21
nighttime incontinence episodes | -0.2 (0.0) | -0.1 (0.0) | -0.2 (0.1) | -0.2 (0.1)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.630, ANCOVA — P-value is from a rank ANCOVA analysis stratified by geographic region; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = 0.1, 95% CI 2-sided [0.0 to 0.2], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.1 — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Dry (Incontinence-Free) Days Per 7 Days
Description: The mean number of dry days was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. An incontinence episode is defined as an episode with any involuntary loss of urine.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Dry Days
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 73 | 19 | 21
Dry Days | 1.7 (0.3) | 1.3 (0.3) | 1.5 (0.8) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.563, ANCOVA — P-value is from a rank ANCOVA analysis stratified by geographic region; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.3], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-1.6 to 1.9], Standard Error of Mean 0.8 — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Dry (Incontinence-Free) Nighttimes Per 7 Days
Description: The mean number of dry nights was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. An incontinence episode is defined as an episode with any involuntary loss of urine.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Dry Nights
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 73 | 19 | 21
Dry Nights | 0.7 (0.2) | 0.4 (0.2) | -0.1 (0.4) | 0.4 (0.4)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.770, ANCOVA — P-value is from a rank ANCOVA analysis stratified by geographic region; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.3], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = 0.5, 95% CI 2-sided [-0.4 to 1.3], Standard Error of Mean 0.4 — [estimate comment as in outcome 1, analysis 2]

8. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Micturitions Per 24 Hours
Description: The mean number of micturitions was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. A micturition is any voluntary urination, excluding episodes of incontinence.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 73 | 19 | 21
micturitions | -0.8 (0.2) | -1.1 (0.2) | -0.6 (0.5) | -0.4 (0.4)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.303, ANCOVA — From an ANCOVA model including treatment, geographic region & gender as fixed effects & the baseline value as a covariate; Adjusted Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.2], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = 0.1, 95% CI 2-sided [-0.9 to 1.1], Standard Error of Mean 0.5 — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Daytime Micturitions Per 24 Hours
Description: The mean number of micturitions was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. A micturition is any voluntary urination, excluding episodes of incontinence. Daytime is defined as the time between waking up in the morning and going to bed later the same day.
Time Frame: Baseline and week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: daytime micturitions
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 71 | 19 | 21
daytime micturitions | -1.1 (0.2) | -1.2 (0.2) | -0.5 (0.5) | -0.3 (0.5)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.640, ANCOVA; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -0.1, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = 0.3, 95% CI 2-sided [-0.9 to 1.4], Standard Error of Mean 0.6 — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Nighttime Micturitions Per 24 Hours
Description: The mean number of micturitions was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit. A micturition is any voluntary urination, excluding episodes of incontinence. Nighttime is defined as the time between going to bed and waking up the following morning.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nighttime micturitions
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 70 | 71 | 19 | 21
nighttime micturitions | 0.0 (0.1) | -0.1 (0.1) | 0.4 (0.3) | 0.1 (0.3)
Statistical Analysis 1: Comparison: Placebo Children vs Solifenacin Succinate Suspension Children; Test type: Superiority or Other; p = 0.846, ANCOVA — P-value is from a rank ANCOVA analysis stratified by geographic region; [statistical method as in outcome 2, analysis 1]; Adjusted Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = -0.2, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.4 — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Grade 3 or 4 Urgency Episodes Per 24 Hours in Adolescents
Description: Adolescent participants were asked to record the degree of urgency associated with each micturition and incontinence episode according to the Patient Perception of Intensity of Urgency Scale (PPIUS) scale (0 - no urgency, 1 - mild urgency, 2 - moderate urgency, 3 - severe urgency, 4 - urge incontinence). The mean number of grade 3 or 4 urgency episodes was determined using using diary data recorded by the participant in the 7 days prior to baseline visit and end of treatment visit.
Time Frame: Baseline and Week 12
Population: The study analysis population for this endpoint consisted of the FAS including participants for whom data were available (adolescents only). Missing values at EoT were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 19 | 20
urgency episodes | -0.7 (0.5) | -1.0 (0.5)
Statistical Analysis 1: Comparison: Placebo Adolescents vs Solifenacin Succinate Suspension Adolescents; Test type: Superiority or Other; Adjusted Mean Difference = -0.3, 95% CI 2-sided [-1.4 to 0.8], Standard Error of Mean 0.5 — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Maximum Concentration (Cmax) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment. Cmax could not be calculated for 2 children and 1 adolescent in the Pharmacokinetic Analysis Set (PKAS).
Time Frame: Week 12/Day 84 (within 3 hours before dosing, 1-3 hours, 4-5 hours, 7-10 hours after dosing) and one sample at Visit 8/Day 87 (2-3 days after last dose intake).
Population: The study analysis population for this endpoint consisted of the PKAS. The PKAS consisted of the subset of the Safety Analysis Set (SAF) for which plasma concentration data were available to facilitate derivation of at least 1 pharmacokinetic parameter and for whom the time of last dose prior to sampling was known.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Children PED 5: Children aged 5 to 11 years of age who received Pediatric Equivalent Dose (PED) 5.0 mg solifenacin succinate suspension
- Children PED 7.5: Children aged 5 to 11 years of age who received Pediatric Equivalent Dose (PED) 7.5 mg solifenacin succinate suspension
- Adolescents PED 7.5: Adolescents aged 12 to 17 years of age who received Pediatric Equivalent Dose (PED) 7.5 mg solifenacin succinate suspension
- Children PED 10: Children aged 5 to 11 years of age who received Pediatric Equivalent Dose (PED) 10 mg solifenacin succinate suspension
- Adolescents PED 10: Adolescents aged 12 to 17 years of age who received Pediatric Equivalent Dose (PED) 10 mg solifenacin succinate suspension
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 6 | 12 | 1 | 46 | 16
ng/mL | 16.67 (4.593) | 26.24 (6.617) | 17.08 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had Cmax measured. | 33.48 (11.93) | 42.85 (21.44)

13. Secondary Outcome: Time to Attain Maximum Concentration (Tmax) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment. Tmax could not be calculated for 2 children and 1 adolescent in the PKAS.
Time Frame: as for outcome 12
Population: The study analysis population for this endpoint consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 6 | 12 | 1 | 46 | 16
hours | 2.933 (0.5354) | 3.175 (0.561) | 2.8 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had Tmax measured. | 2.874 (0.5268) | 2.85 (0.4733)

14. Secondary Outcome: Plasma Concentration Before Drug Administration (Ctrough) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment. Ctrough could not be calculated for 2 children and 1 adolescent in the PKAS.
Time Frame: as for outcome 12
Population: The study analysis population for this endpoint consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 6 | 12 | 1 | 46 | 16
ng/mL | 9.534 (3.083) | 16.1 (4.951) | 8.828 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had Ctrough measured. | 19.05 (8.7) | 27.94 (16.76)

15. Secondary Outcome: Area Under the Plasma Concentration - Time to Curve (AUC) for a Dose Interval (AUCtau) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment.
Time Frame: as for outcome 12
Population: The study analysis population for this endpoint consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 8 | 12 | 1 | 46 | 17
ng*h/mL | 298.7 (80.35) | 452.8 (112.6) | 269.2 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had AUCtau measured. | 560 (216.8) | 745.7 (411)

16. Secondary Outcome: Apparent Terminal Elimination Half-Life (T1/2) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment.
Time Frame: as for outcome 12
Population: The study analysis population for this endpoint consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 8 | 12 | 1 | 46 | 17
hours | 27.3 (5.486) | 30.98 (7.147) | 24.84 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had t1/2 measured. | 26.85 (7.475) | 41.27 (17.44)

17. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment.
Time Frame: as for outcome 12
Population: The study analysis population for this endpoint consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 8 | 12 | 1 | 46 | 17
L/h | 6.968 (2.129) | 7.608 (1.782) | 14.56 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had CL/F measured. | 8.773 (3.763) | 11.3 (7.294)

18. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Solifenacin
Description: Pharmacokinetic sampling was performed at steady state at the end of treatment.
Time Frame: as for outcome 12
Population: The study analysis population for this endpoint consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Children PED 5 | Children PED 7.5 | Adolescents PED 7.5 | Children PED 10 | Adolescents PED 10
Number analyzed (Participants) | 8 | 12 | 1 | 46 | 17
L | 272.4 (96.84) | 329.5 (63.32) | 521.9 (NA) — Standard deviation is not applicable, only one adolescent participant received PED 7.5 that had Vz/F measured. | 315.7 (96.23) | 561.7 (181.7)

19. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A treatment emergent adverse event (TEAE) was defined as an AE that occurred after the first dose of study drug and within 7 days after last dose of study medication.
Time Frame: From the first dose of study drug until 7 days after last dose of study medication (13 weeks).
Population: The study analysis for this endpoint consisted of the Safety Analysis Set (SAF), the SAF consisted of all patients who received at least 1 dose of double-blind study medication and for whom any safety data were reported after first dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 73 | 73 | 19 | 22
participants
  Any TEAE | 45 | 44 | 12 | 9
  Drug Related TEAEs | 9 | 14 | 2 | 3
  Deaths | 0 | 0 | 0 | 0
  Serious TEAEs | 2 | 2 | 1 | 1
  Drug-related Serious TEAEs | 1 | 0 | 0 | 0
  TEAEs Leading to Discontinuation | 1 | 6 | 2 | 2
  Drug-related TEAEs Leading to Permanent Discont. | 1 | 3 | 1 | 1

20. Secondary Outcome: Change From Baseline in Post Void Residual (PVR) Volume
Description: Post Void Residual (PVR) Volume was assessed by ultrasonography or bladder scan.
Time Frame: Baseline and Week 12
Population: The study analysis population for this endpoint consisted of the SAF.
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Number analyzed (Participants) | 73 | 73 | 19 | 22
mL | 0.07 (7.28) | -0.99 (6.45) | -3.58 (4.72) | 0.95 (9.85)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 7 days after last dose of study medication (13 weeks).
Groups:
- Placebo Children: Children aged 5 to 11 years received matching placebo oral suspension once a day for 12 weeks.
- Solifenacin Succinate Suspension Children: Children aged 5 to 11 years received solifenacin succinate suspension once a day for 12 weeks.
- Placebo Adolescents: Adolescents aged 12 to 17 years received matching placebo oral suspension once a day for 12 weeks.
- Solifenacin Succinate Suspension Adolescents: Adolescents aged 12 to 17 years received solifenacin succinate suspension once a day for 12 weeks.
Arm/Group | Placebo Children | Solifenacin Succinate Suspension Children | Placebo Adolescents | Solifenacin Succinate Suspension Adolescents
Serious Adverse Events (participants affected / at risk) | 2/73 | 2/73 | 1/19 | 1/22
Other Adverse Events (participants affected / at risk) | 26/73 | 28/73 | 12/19 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Children (N=73) | Solifenacin Succinate Suspension Children (N=73) | Placebo Adolescents (N=19) | Solifenacin Succinate Suspension Adolescents (N=22)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frontal lobe epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Children (N=73) | Solifenacin Succinate Suspension Children (N=73) | Placebo Adolescents (N=19) | Solifenacin Succinate Suspension Adolescents (N=22)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (8) | 6 (6) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 5 (7) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 90 days prior to publication for review and comment. Sponsor may delay the publication temporarily to seek patent protection or permanently withhold the publication.